CLINICAL TRIAL: NCT07389486
Title: A Comparative Study of Continuous vs. Intermittent Real-time fMRI Neurofeedback in Regulating Anterior Insula Activity
Brief Title: Continuous vs. Intermittent Rt-fMRI Neurofeedback Training of the Anterior Insula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-104
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Real-time neurofeedback; Anterior insula; Feedback types; Interoceptive processing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent neurofeedback training (Experimental): Subjects in the intermittent neurofeedback training group are instructed to regulate their anterior insula activity based on the visual neurofeedback after each regulation block. This intermittent neurofeedback is based on averaged activity of the anterior insula during the regulation block.
  Interventions: Procedure: real-time fMRI neurofeedback training procedure
- Intermittent sham control (Sham Comparator): Subjects in the sham control group receive the same instruction but perform the regulation based on sham neurofeedback from the middle temporal gyrus (a controlled sham region).
  Interventions: Procedure: real-time fMRI sham-controlled neurofeedback training procedure
- Continuous neurofeedback training (Experimental): Subjects in the continuous neurofeedback training group are instructed to regulate their anterior insula activity based on the real-time visual neurofeedback during regulation blocks.
  Interventions: Procedure: real-time fMRI neurofeedback training procedure

INTERVENTIONS:
Procedure: real-time fMRI neurofeedback training procedure — real-time fMRI neurofeedback training procedure running on the Turbo Brain voyager (TBV) 4.2 software (Brain Innovation, Maastricht, The Netherlands)
  Arms: Intermittent neurofeedback training
Procedure: real-time fMRI sham-controlled neurofeedback training procedure — real-time fMRI sham neurofeedback training procedure running on the Turbo Brain voyager (TBV) 4.2 software (Brain Innovation, Maastricht, The Netherlands)
  Arms: Intermittent sham control
Procedure: real-time fMRI neurofeedback training procedure — real-time fMRI neurofeedback training procedure running on the Turbo Brain voyager (TBV) 4.2 software (Brain Innovation, Maastricht, The Netherlands)
  Arms: Continuous neurofeedback training

SUMMARY:
The main aim of this study is to compare the efficacy of intermittent with continuous real-time functional magnetic resonance imaging (fMRI) neurofeedback on anterior insula regulation and associated behavioral changes.

DETAILED DESCRIPTION:
A double-blinded, placebo-controled, between-subject design is employed in this study. A total of 90 healthy subjects will be recruited and randomly assigned into the intermittent experimental group (EG1; N=30), which receives intermittent feedback from the left anterior insula after each block, the control group (CG; N=30) after each block, which receives sham feedback from the middle temporal gyrus (MTG), and the continuous expermiental group (EG2; N=30), which receives real-time feedback from the left anterior insula. Comparisons between the EG1 and the CG are used to validate the efficacy of intermittent neurofeedback and comparisons between the EG2 and the CG are used to determine the better neurofeedback type (intermittent vs. continuous).

The neurofeedback training task consists of 4 training sessions with real-time feedback and 1 transfer session without feedback. Each session comprises 5 regulation blocks and 5 rest blocks. At the end of each block, participants are presented with pain-related images and asked to rate their level of pain empathy, which was used to determine the effects of neurofeedback training on empathic responses. A heartbeat detection task is performed pre- and post-training to measure interoceptive accuracy changes induced by neurofeedback training. A functional localizer task (heartbeat counting task) before training was used to localise the anterior insula. Personality traits of subjects are assessed using validated Chinese version questionnaires, including the Toronto Alexithymia Scale (TAS), Multidimensional Assessment of Interoceptive Awareness (MAIA), Bermond-Vorst Alexithymia Questionnaire (BVAQ),Interoceptive Confusion Questionnaire (ICQ), Beck Depression Inventory (BDI), State-Trait Anxiety Inventory (STAI), Autism Spectrum Quotient (ASQ), Interpersonal Reactivity Index (IRI), and Cognitive Flexibility Inventory (CFI). Subjects are asked to complete Positive and Negative Affect Schedule (PANAS) twice before and after the neurofeedback training task to measure mood changes.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

History of brain injury medical or mental illness

Contraindication to MRI scanning (e.g., metal implants, claustrophobia or other --conditions that make them inappropriate for MRI scanning)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals whose self-identified gender is consistent with their biological sex.
Enrollment: 90 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
Neural activity of the anterior insula based on blood oxygen level-dependent (BOLD) signal | 1 hour
  The anterior insula activity induced during the regulation block compared to the baseline block.
Pain empathy ratings scores | 1 hour
  Subjects were required to rate their empathic feeling towards painful pictures on a Likert Scale ranging from 1-9 (1 = not at all and 9 = very painful) before and after neurofeedback training.

SECONDARY OUTCOMES:
Confidence rating scores of interoceptive sensitivity | 1 hour
  Subjects are asked to rate to what extent they can feel their heartbeat based on a Likert Scale ranging from 1-9 (1 = very low and 9 = very high)
Interoceptive accuracy | 10 minutes
  1/N Σ(1-(|actual heartbeats--reported heartbeats|) / actual heartbeats). N indicates the number of recording blocks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China